CLINICAL TRIAL: NCT00148395
Title: Randomized Phase III-Study in Stage IIIb and IV Non-Small-Cell Lung Cancer. Sequential Single-Agent vs. Double-Agent vs. Triple-Agent Therapy.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Aktion Bronchialkarzinom e.V. (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NSCLC 06/2001
Record Dates: First submitted 2005-09-07; First posted 2005-09-08 (Estimated); Last update posted 2008-04-22 (Estimated); Status verified 2008-04

CONDITIONS: Non-Small-Cell Lung Carcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Gemcitabine; Vinorelbine; Carboplatin; Cisplatin; Mitomycin; Ifosfamide

INTERVENTIONS:
Drug: Gemcitabine
Drug: Navelbine
Drug: Carboplatin
Drug: Cisplatin
Drug: Mitomycin
Drug: Ifosfamide

SUMMARY:
This study wants to assess different intensive therapy sequences for the treatment of non-small-cell lung cancer.

It claims less on the efficacy of different chemotherapy combinations, than more on the comparison of different strategies of sequential single-agent, sequential double-agent or sequential triple-agent therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Histological verified non-small cell lung cancer. Cytological diagnosis is accepted for doubtless results.
2. Present stage IIIb with malignant pleural effusion or stage IV disease. Tumor dissemination should not be irradiable in one field
3. Age between 18 and 75 years
4. Karnofsky index 70 - 100%
5. Measurable or evaluable tumor parameter
6. No prior chemotherapy for NSCLC
7. Sufficient hematological parameter before start of therapy (leucocytes > 3.500/µl and platelets > 100.000/µl).
8. Sufficient liver function (bilirubin < 1,6mg/dl)
9. Sufficient renal function (creatinine < 1,5mg/dl and clearance > 60ml/min)
10. Minimal estimated life expectancy > 3 months
11. Written informed consent for study attendance
12. Patient accessibility for therapy and follow up
13. No attendance to an other study

Exclusion Criteria:

1. Small-cell lung cancer oder tumors with small-cell fractions
2. Local advanced irradiable stage III
3. Previous chemotherapy because of other diseases, not longer than 3 years ago
4. Simultaneous radiation of all present tumor manifestations
5. Simultaneous or not longer than 3 years ago secondary malignancy, except carcinoma in situ of the cervix or dermal cancer, others than melanoma
6. Respiratory insufficiency
7. Heart insufficiency NYHA III and IV
8. Peripheral arteriosclerosis stage III and IV
9. Neurological and psychiatric diseases, which affect understanding of the study concept and the possibility to keep conditions of the protocol
10. Pregnancy, breastfeeding or not ensured contraception
11. HIV-infection
12. Active hepatitis B and C
13. Manifest infectious diseases before start of therapy
14. Minimal estimated life expectancy < 3 months
15. No written informed consent of the patient for study attendance and storage and disclosure of disease data according to the protocol

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280
Dates: Start 2002-06; Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Overall survival

SECONDARY OUTCOMES:
Event-free survival
Quality of live

CONTACTS AND LOCATIONS:
Overall Officials: Martin Wolf, MD, Study Chair — Klinikum Kassel GmbH
Locations (1):
- Klinikum Kassel GmbH, Kassel, Germany